CLINICAL TRIAL: NCT03703674
Title: Granulocyte Colony Stimulating Factor in Alcoholic Hepatitis
Brief Title: GCSF in Alcoholic Hepatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCSF IN ALCOHOLIC HEPATITIS
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Therapy (Active Comparator): Drug: standard medical therapy Standard medical therapy involves primary treatment and normal hospital nutrition (1800 to 2000 kcal per day). Diuretics, sodium restriction and albumin for treatment of ascites or fresh frozen plasma for coagulopathy or antibiotics for any focus of infection as spontaneous bacterial peritonitis (SBP), pneumonia, cellulitis, and urinary tract infection as indicated.
  Interventions: Drug: GCSF
- G-CSF + Standard Medical Therapy (Experimental): Drug: standard medical therapy Standard medical therapy involves primary treatment and normal hospital nutrition (1800 to 2000 kcal per day). Diuretics, sodium restriction and albumin for treatment of ascites or fresh frozen plasma for coagulopathy or antibiotics for any focus of infection as spontaneous bacterial peritonitis (SBP), pneumonia, cellulitis, and urinary tract infection as indicated.
  Drug: G-CSF G-CSF- 5 μg/Kg s.c every 12 hours for 5 consecutive days
  Interventions: Drug: GCSF

INTERVENTIONS:
Drug: GCSF — Granulocyte-colony stimulating factors (G-CSF)

SUMMARY:
Alcoholic hepatitis is related to very high mortality rate. About 40% of the patients are died within first 6 months after the detection of the clinical syndrome. Therefore, it is very essential for proper diagnosis and early treatment. In response to acute or chronic liver damage, bone marrow derived stem cells can spontaneously populate liver and differentiate into hepatic cells. Animal and human studies suggested that injured hepatocyte may be replaced by pluripotent bone marrow cells. However, this hepatocyte repopulation is highly dependent on varieties of liver injury and therapeutic conditions. The studies has suggested Granulocyte-colony stimulating factors (G-CSF) can regenerate hepatocyte by fusing with hematopoietic cells, thereby enhancing the liver histology and survival rate.

G-CSF is a cytokine capable to regulate a number of functions in neutrophils. In three recent studies mobilization of bone marrow stem cells induced by G-CSF was observed in patients with alcoholic hepatitis. In two of this studies there was a survival benefit with the use of G-CSF.

Therefore we plan to study the safety and efficacy of G-CSF in the patients with alcoholic hepatitis.

DETAILED DESCRIPTION:
Detailed Description:

Patients with severe alcoholic hepatitis, admitted to Department of Hepatology PGIMER, Chandigarh will be included in the study.

METHODS

This will be an open label trial. A randomization code is generated by random number table. The patients will be randomized to receive standard medical therapy (SMT) only as control and therapy of G-CSF as case. There will be one control and one case as below:

1) SMT (control) 2) G-CSF (case): G-CSF 5 mcg/kg every 12 hourly for consecutive 5 days This will be a single time therapy. Patients will be admitted in the department of hepatology and will be assessed everyday clinically as well as by laboratory tests during therapy to assess safety and effects of treatment.

1. Total leukocytes count will be assessed daily.
2. Circulating CD 34 positive cells will be measured on day 0 and 6 of G-CSF therapy.
3. In addition, ultrasonography will be performed at day 1 and 6 in order to evaluate difference in spleen size and portal vein flow.
4. Biochemical, coagulation, and hematological parameters (Liver function tests, Renal Function Tests, Prothrombin Time, International Normalised Ratio, etc.) will be monitored periodically, daily for 1 week, then weekly for 1month and monthly for three month.

All patients will be followed at weekly interval for 1 month and then monthly for 3 months.

Outcome:

Primary Objectives:

Survival at 3 months

Secondary Objectives:

Mobilisation of CD34 positive cells in peripheral blood.Clinical/biochemical improvement in liver function profile.Improvement in prognostic scores-Maddrey's Discriminant function, MELD score, and Child score.

Safety and efficacy of G-CSF in alcoholic hepatitis

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic hepatitis patients:

  1. More than 10 years of heavy alcohol consumption (mean intake ≈ 100 g/day).
  2. Elevated aspartate aminotransferase level (but <500 IU per millilitre) and Ratio ofAST/ALT≥2 times
  3. Elevated serum total bilirubin level ≥ 5 mgdL (86 μmol/L)
  4. Elevated INR(≥1.5) and
  5. Neutrophilia. Patient with Maddrey's DF of ≥ 32 will be included in the study, with or without biopsy.

Exclusion Criteria:

* 1. Age < 18 and > 75 years 2. Hepatocellular carcinoma or portal vein thrombosis 3. Refusal to participate in the study 4. Serum creatinine>1.0 mg% 5. Hepatic encephalopathy- grade 3 or 4 6. Upper gastrointestinal bleed in last ten days 7. Uncontrolled bacterial infection 8. Human immunodeficiency virus, Hepatitis B virus, Hepatitis C virus seropositivity, Autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency 9. Pregnancy 10. Glucocorticoid treatment 11. Significant co-morbidity 12. Previous known hypersensitivity to G-CSF

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-19 (Actual); Primary Completion 2020-11-18 (Estimated); Study Completion 2020-11-18 (Estimated)

PRIMARY OUTCOMES:
Survival at 3 months | 90 DAYS

SECONDARY OUTCOMES:
Mobilisation of CD34 positive cells in peripheral blood. | 6 DAYS
Improvement in MELD score | 90 DAYS
Improvement in Maddrey's Discriminant Function. | 90 Days
Improvement in Child Turcotte Pugh score. | 90 Days
Number of participants with treatment-related adverse events in the different groups. | 90 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No